CLINICAL TRIAL: NCT06584097
Title: COMparative Performance of General Purpose Models for Propofol And REmifentanil in Neurosurgical Patients Admitted to the Intensive Care Unit
Brief Title: COMparative Performance of General Purpose Models
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: COMPARE ICU
Record Dates: First submitted 2024-07-10; First posted 2024-09-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neurosurgical Patients
Keywords: Neuroanesthesia; total intravenous anesthesia; target controlled infusion; PKPD modelling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To compare the performance of the Eleveld models for propofol and remifentanil on neurosurgery patients admitted to intensive care with their intraoperative performance.

DETAILED DESCRIPTION:
Despite the widespread adoption of Target Controlled Infusion (TCI) models in modern clinical anesthesia practice, much less attention has been paid in the literature to their potential applications in the Intensive Care Unit (ICU) setting. Few studies have been published so far to evaluate the performance of TCI pumps for sedatives and other drugs (e.g., antibiotics) in Intensive Care. Further data is needed regarding the use of TCI for the long-term infusion of these drugs in the ICU after surgery, and the quantitative relationship between generalized pharmacokinetic/pharmacodynamic models for propofol and remifentanil (the Eleveld models) has yet to be evaluated in this specific population. This study is an observational study with the aim of clarifying the predictive performance of the TCI models for the administration of propofol and remifentanil in a cohort of intensive care patients admitted after neurosurgery and compare it to the intraoperative performance, which can be taken as benchmark.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective neurosurgical procedures with an expected sedation after surgery of > 12 hours • Requirement for an arterial line

Exclusion Criteria:

* Pregnancy

  * Known sensitivity or allergy to propofol or remifentanil
  * Patient participating in research for which a period of exclusion is currently required by other study protocol, ethical committee or health authority.
  * Age < 18 years old
  * Patients subjected to infusion of propofol and/or remifentanil not delivered through TCI pumps before the inclusion
  * Patients exposed to other sedatives (benzodiazepines, volatile anesthetics, quetiapine) before the inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients undergoing elective neurosurgical procedures with an expected sedation after surgery of > 12 hours
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MdAPE difference for propofol | october 2024
  The difference in MdAPE will be measured when comparing the model performance for propofol in the ICU to the intraoperative phase.
MdAPE difference for remifentanil | october 2024
  The difference in MdAPE will be measured when comparing the model performance for remifentanil in the ICU to the intraoperative phase.

SECONDARY OUTCOMES:
Propofol and remifentanil metabolites | october 2024
  Metabolites of propofol and remifentanil (4-hydroxy propofol and remifentanil acid) during infusion
BIS profile | october 2024
  Bispectral index monitor profile during infusion (min = 0, max = 100)
NOL profile | Oct 2024
  NOL (Nociceptive Level) value (min = 0, max = 100)
RASS | october 2024
  RASS measurements during infusion (min = -5, max = +4).

CONTACTS AND LOCATIONS:
Overall Officials: Michele Introna, M.d., Principal Investigator — Fondazione IRCCS Istituto Neurologico C. Besta
Locations (2):
- Italy (2):
  - Foundation IRCCS Carlo Besta Neurological Institute, Milan, Italy
  - Fondazione IRCCS Istituto Neurologico C. Besta, Milan, Milano

IPD SHARING:
Plan to Share IPD: Yes
Propofol and remifentanil pharmacokinetic and pharmacodynamic data.